CLINICAL TRIAL: NCT04032613
Title: Breaking Down Care Process and Patient-level Barriers to Arteriovenous Access Creation Prior to Hemodialysis Initiation: a Pilot Study
Brief Title: Breaking Down Care Process and Patient-level Barriers to Arteriovenous Access Creation Prior to Hemodialysis Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Geisinger Clinic (Other); Duke University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-1912; 1R21DK116115 (NIH)
Record Dates: First submitted 2019-06-26; First posted 2019-07-25 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-08

CONDITIONS: Chronic Kidney Disease; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hemodialysis; Vascular access; Arteriovenous; Dialysis; End Stage Renal Disease; Patient-reported outcomes; Feasibility; Care process; Patient education; Health system navigation; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This study uses a pre-intervention / post-intervention design to assess outcomes. The study measures the pre-intervention to post-intervention changes in participant: 1) vascular access knowledge, and 2) confidence in navigating dialysis vascular access care process steps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascular access quality improvement program participants (Experimental): All participants enrolled in the study who are involved in the Vascular Access Navigation and Education Quality Improvement Program.
  Interventions: Other: Vascular Access Navigation and Education Quality Improvement Program

INTERVENTIONS:
Other: Vascular Access Navigation and Education Quality Improvement Program — A Vascular Access Navigation and Education Quality Improvement Program implemented in the Geisinger Danville, PA chronic kidney disease clinic. Participants complete questionnaires to assess their vascular access care knowledge and confidence before and after the implementation of the quality improvement program.

SUMMARY:
More than 80% of individuals in the U.S. start maintenance hemodialysis (HD) with a central venous catheter, despite substantial evidence that starting HD with an arteriovenous (AV) access improves quality of life, lowers mortality, and decreases healthcare costs. Health system- and patient-level barriers contribute to low rates of AV access creation prior to HD initiation. Evidence-based, pre-dialysis interventions to improve these low rates and associated clinical outcomes are lacking.

A Vascular Access Navigation and Education Quality Improvement Program will be implemented in the Geisinger Danville, PA chronic kidney disease clinic. Individuals who choose to participate in a research sub-study of the program will complete questionnaires to assess their vascular access care knowledge and confidence before and after participation in the quality improvement program.

ELIGIBILITY:
Inclusion Criteria

Patients:

* Receive care at the Geisinger Danville Nephrology Clinic
* Age ≥ 18 years
* eGFR ≤ 25 mL/min/1.73 m and 2-year kidney failure risk score >10% based on kidney failure risk equation, or nephrologist recommendation for vascular access
* Participation in the Vascular Access Navigation and Education Quality Improvement Program

Providers: Professional involved in dialysis vascular access care (e.g., nephrologist, surgeon, kidney disease clinic nurse, etc.) at Geisinger in Danville, PA

Exclusion Criteria

Patients:

* Too far into the vascular access creation process to benefit from the intervention (e.g. completed vascular access surgery appointment or has a surgery appointment scheduled within the next 4 weeks),
* Inability to consent, or
* Inability to complete interviews in English

Providers: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Flythe, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Jamie Green, MD, MS, Principal Investigator — Geisinger Clinic; Ebony Boulware, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Geisinger Danville Nephrology Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data generated in this study are protected under data use agreements among Geisinger, Duke University, and the University of North Carolina at Chapel Hill. We cannot directly share the source data without written approval from these institutions. If scientists are interested in accessing de-identified study data, we will work with all institutions to obtain the necessary data use agreement modifications.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication, pending data use agreement modifications.
Access Criteria: Principal Investigators will review all requests for data, per data use agreement modifications.

REFERENCES:
- [Derived] Flythe JE, Narendra JH, Yule C, Manivannan S, Murphy S, Lee SD, Strigo TS, Peskoe S, Pendergast JF, Boulware LE, Green JA. Targeting Patient and Health System Barriers To Improve Rates of Hemodialysis Initiation with an Arteriovenous Access. Kidney360. 2021 Feb 26;2(4):708-720. doi: 10.34067/KID.0007812020. eCollection 2021 Apr 29. PMID 35373037

RESULTS

PARTICIPANT FLOW:
Groups:
- Vascular Access QI Program Patient Participants: All patient participants enrolled in the study who are involved in the Vascular Access Navigation and Education Quality Improvement (QI) Program.
  Vascular Access Navigation and Education Quality Improvement Program: A Vascular Access Navigation and Education Quality Improvement Program implemented in the Geisinger Danville, PA chronic kidney disease clinic. Participants complete questionnaires to assess their vascular access care knowledge and confidence before and after the implementation of the quality improvement program.
- Vascular Access QI Program Provider/Personnel Participants: All provider/personnel participants enrolled in the study who are involved in the Vascular Access Navigation and Education Quality Improvement Program.
  Vascular Access Navigation and Education Quality Improvement Program: A Vascular Access Navigation and Education Quality Improvement Program implemented in the Geisinger Danville, PA chronic kidney disease clinic. Participants complete questionnaires to assess their vascular access care knowledge and confidence before and after the implementation of the quality improvement program.
Period: Overall Study
Arm/Group | Vascular Access QI Program Patient Participants | Vascular Access QI Program Provider/Personnel Participants
Started | 21 | 25
Completed | 16 | 23
Not Completed | 5 | 2
Not completed — Did not complete post-program assessment | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Vascular Access QI Program Patient Participants: All patient participants enrolled in the study who are involved in the Vascular Access Navigation and Education Quality Improvement Program.
  Vascular Access Navigation and Education Quality Improvement Program: A Vascular Access Navigation and Education Quality Improvement Program implemented in the Geisinger Danville, PA chronic kidney disease clinic. Participants complete questionnaires to assess their vascular access care knowledge and confidence before and after the implementation of the quality improvement program.
- Total: Total of all reporting groups
Arm/Group | Vascular Access QI Program Patient Participants | Vascular Access QI Program Provider/Personnel Participants | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (15.2) | 39.6 (6.9) | 50.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 22 | 43
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Mean Scores of a Questionnaire Evaluating Patient Confidence in Navigating Vascular Access Care Pre- to Post-program Implementation
Description: Patient confidence in ability to navigate the vascular access creation process. Measured using 3 team-developed confidence questions (score range: 1-10). Higher scores reflect higher confidence in navigating vascular access care.
Time Frame: Pre- and post-intervention, a total of up to 7 months
Population: All Vascular Access QI program patient participants enrolled in the study who completed both the pre- and post-program evaluation questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vascular Access QI Program Patient Participants
Number analyzed (Participants) | 16
score on a scale
  Pre-program score mean | 8.0 (1.3)
  Post-program score mean | 8.7 (1.3)
Statistical Analysis 1: Comparison: Vascular Access QI Program Patient Participants; Test type: Other — Paired sample t-test; p = 0.20, Paired sample t-test — Statistically significant p-value is <0.05

2. Primary Outcome: Mean Scores of a Questionnaire Evaluating Patient Confidence in Self-managing Kidney Disease Pre- to Post-program Implementation
Description: Patient confidence in ability to self-manage kidney disease. Measured using a modified version of the 8-item Perceived Kidney Disease Self-Management Scale (score range: 8-40). Higher scores reflect higher confidence in self-management of patient's kidney disease.
Time Frame: Pre- and post-intervention, a total of up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vascular Access QI Program Patient Participants
Number analyzed (Participants) | 16
score on a scale
  Pre-program score mean | 28.1 (4.1)
  Post-program score mean | 30.8 (5.3)
Statistical Analysis 1: Comparison: Vascular Access QI Program Patient Participants; Test type: Other — Paired sample t-test; p = 0.05, Paired sample t-test — Statistically significant p-value is <0.05

3. Primary Outcome: Mean Scores of a Questionnaire Evaluating Patient Vascular Access Knowledge Pre- to Post-program Implementation
Description: Patient vascular access care knowledge. Measured using 8 team-developed knowledge questions (score range: 0-10). Higher scores reflect higher knowledge of vascular access.
Time Frame: Pre- and post-intervention, a total of up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vascular Access QI Program Patient Participants
Number analyzed (Participants) | 16
score on a scale
  Pre-program score mean | 4.9 (2.8)
  Post-program score mean | 6.9 (1.9)
Statistical Analysis 1: Comparison: Vascular Access QI Program Patient Participants; Test type: Other — Paired sample t-test; p = 0.004, Paired sample t-test — Statistically significant p-value is <0.05

4. Primary Outcome: Mean Scores of a Questionnaire Evaluating Provider Confidence Supporting Patients Through the Vascular Access Care Process Pre- to Post-program Implementation
Description: Provider confidence in ability to help patients navigate the vascular access creation process. Measured using 11 team-developed confidence questions (score range: 1-10). Higher scores reflect higher confidence supporting patients through the vascular access care process.
Time Frame: Pre- and post-intervention, a total of up to 7 months
Population: All Vascular Access QI program provider & personnel participants enrolled in the study who completed both the pre- and post-program evaluation questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vascular Access QI Program Provider/Personnel Participants
Number analyzed (Participants) | 23
score on a scale
  Pre-program score mean | 7.5 (0.9)
  Post-program score mean | 7.8 (0.8)
Statistical Analysis 1: Comparison: Vascular Access QI Program Provider/Personnel Participants; Test type: Other — Paired sample t-test; p = 0.14, Paired sample t-test — Statistically significant p-value is <0.05

ADVERSE EVENTS:
Time Frame: From the time informed consent is obtained to study participation end, an approximate total of 7 months.
Arm/Group | Vascular Access QI Program Patient Participants | Vascular Access QI Program Provider/Personnel Participants
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 0/21 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04032613/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04032613/SAP_001.pdf